CLINICAL TRIAL: NCT05718232
Title: Stereotactic Body Radiation Therapy Plus Lenvatinib and Transarterial Chemoembolization for Advanced Primary Hepatocellular Carcinoma: A Phase 3, Multicentric, Randomized Controlled Trial
Brief Title: SBRT Plus Lenvatinib and TACE for Advanced Primary HCC: A Phase 3 Trial (SEARCH)
Acronym: SEARCH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCC202210
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: SBRT; TACE; Lenvatinib
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT+TACE+Lenvatinib (Experimental): Patients in SBRT+TACE+Lenvatinib group will take oral lenvatinib within 3 days of randomization and receive TACE 1 day after oral administration of lenvatinib. SBRT will begin within 3 weeks after the first TACE.
  Interventions: Drug: Lenvatinib; Procedure: TACE; Radiation: SBRT
- Lenvatinib (Active Comparator): Patients in Lenvatinib group will take oral lenvatinib alone.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be taken within 3 days of randomization (dose: 8 mg qd for patients <60kg, and 12 mg qd for patients ≥ 60kg)
Procedure: TACE — TACE will be performed one day after oral administration of lenvatinib. Either cTACE or DEB-TACE can be used, depending on the condition of each center.
  Arms: SBRT+TACE+Lenvatinib
Radiation: SBRT — SBRT will be given within 3 weeks after the first TACE with linear accelerator-based photon beams. Gross tumor volume is defined as intrahepatic tumor and vascular invasion including a 1-cm margin into the contiguous HCC. Prescription dose will be 4500-5000 cGy in 5-8 fractions.
  Arms: SBRT+TACE+Lenvatinib

SUMMARY:
This is a phase 3, multicentri, randomised, open label study. The purpose is to investigate the safety and efficacy of stereotactic body radiation therapy (SBRT) combined with transarterial chemoembolization (TACE) and lenvatinib (LEN) in the treatment of advanced hepatocellular carcinoma with portal vein tumor thrombus.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old;
2. Patients with primary advanced HCC (in accordance with AASLD2018 guidelines for the diagnosis of HCC), without any previous treatment;
3. There is at least one measurable lesion in the liver according to mRECIST criteria, single tumor ≤ 10.0 cm or multiple tumors and tumor burden ≤50% , with portal vein tumor embolus;
4. ECOG score 0-1;
5. Child-Pugh class A;
6. Expected survival time ≥ 3 months;
7. Blood, liver and kidney function meet the following conditions: Neutrophil count ≥ 1.5 × 10 9 /L; Platelet count ≥ 60 × 10 9 /L; Hemoglobin ≥ 90 g/L; Serum albumin ≥ 30 g/L; Bilirubin ≤ 50 umol/L; AST, ALT ≤ 5 times the upper limit of normal, ALP ≤ 4 times the upper limit of normal; Prolongation of prothrombin time not to exceed the upper limit of normal by 6 seconds; Creatinine ≤ 1.5 times the upper limit of normal.

Exclusion Criteria:

1. Extrahepatic metastases;
2. Previous history of liver or adjacent tissue radiation;
3. Previous history of hepatic encephalopathy, refractory ascites or gastric esophageal varices;
4. There are contraindications to TACE treatment, such as portosystemic shunt, liver flow ablation, significant atherosclerosis;
5. Hypersensitivity to intravenous contrast agents;
6. Pregnant or lactating women or subjects with family planning within two years;
7. With HIV, syphilis infection;
8. Accompanied by other malignant tumors or suffering from other malignancies within 5 years before enrollment;
9. Allogeneic organ transplant recipients;
10. Severe dysfunction of heart and kidney or other organs;
11. Active severe infection > grade 2 (NCI-CTC version 5);
12. Suffering from mental and psychological diseases may affect informed consent;
13. Unable to take oral medication;
14. Participated in other drug clinical trials within 12 months before enrollment;
15. Active gastric or duodenal ulcers within 3 months before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from first treatment to death, regardless of disease recurrence.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the first treatment to progression or death.
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the percentage of patients who have achieved complete response (CR) or partial response (PR), as measured by modified Response Evaluation Criteria in Solid Tumors (mRECIST) criteria.
Disease Control Rate (DCR) | Up to 2 years
  DCR is defined as the percentage of patients who have achieved CR, PR or stable disease(SD), as measured by mRECIST criteria.
Incidence of Adverse Events (AE) | Up to 2 years
  Incidence of AE is defined as the percentage of patients who suffer adverse events from the first treatment to last follow-up, assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Time to Progression （TTP） | Up to 2 years
  TTP is defined as the time from the first treatment to progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, Ph.D., Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peng Z, Fan W, Zhu B, Wang G, Sun J, Xiao C, Huang F, Tang R, Cheng Y, Huang Z, Liang Y, Fan H, Qiao L, Li F, Zhuang W, Peng B, Wang J, Li J, Kuang M. Lenvatinib Combined With Transarterial Chemoembolization as First-Line Treatment for Advanced Hepatocellular Carcinoma: A Phase III, Randomized Clinical Trial (LAUNCH). J Clin Oncol. 2023 Jan 1;41(1):117-127. doi: 10.1200/JCO.22.00392. Epub 2022 Aug 3. PMID 35921605
- [Background] Abulimiti M, Li Z, Wang H, Apiziaji P, Abulimiti Y, Tan Y. Combination Intensity-Modulated Radiotherapy and Sorafenib Improves Outcomes in Hepatocellular Carcinoma with Portal Vein Tumor Thrombosis. J Oncol. 2021 Dec 3;2021:9943683. doi: 10.1155/2021/9943683. eCollection 2021. PMID 34899910
- [Background] Yoon SM, Ryoo BY, Lee SJ, Kim JH, Shin JH, An JH, Lee HC, Lim YS. Efficacy and Safety of Transarterial Chemoembolization Plus External Beam Radiotherapy vs Sorafenib in Hepatocellular Carcinoma With Macroscopic Vascular Invasion: A Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):661-669. doi: 10.1001/jamaoncol.2017.5847. PMID 29543938